CLINICAL TRIAL: NCT02444247
Title: Motivation to Exercise
Acronym: Motiv2Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC400
Record Dates: First submitted 2015-05-07; First posted 2015-05-14 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity; Physical Activity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Exercise vs Sedentary Option (Other): Relative Reinforcing Value of high dose exercise (300 kcal expenditure per session) versus sedentary activity will be determined.
  Interventions: Other: High Dose Exercise (300 kcal); Other: Sedentary Option
- Low Dose Exercise vs Sedentary Option (Other): Relative Reinforcing Value of low dose exercise (150 kcal expenditure per session) versus sedentary activity will be determined.
  Interventions: Other: Low Dose Exercise (150 kcal); Other: Sedentary Option
- No Exercise vs Sedentary Option (Other): Relative Reinforcing Value of no exercise (0 kcal expenditure per session) versus sedentary activity will be determined.
  Interventions: Other: No Exercise (0 kcal); Other: Sedentary Option

INTERVENTIONS:
Other: High Dose Exercise (300 kcal) — Subjects will participate in 3 physical activity sessions per week expending 300 kcal per session and rate their liking of exercise.
  Arms: High Dose Exercise vs Sedentary Option
Other: Low Dose Exercise (150 kcal) — Subjects will participate in 3 physical activity sessions per week expending 150 kcal per session and rate their liking of exercise.
  Arms: Low Dose Exercise vs Sedentary Option
Other: No Exercise (0 kcal) — Subjects will participate in 3 sessions per week expending 0 kcal per session and rate their liking of exercise.
  Arms: No Exercise vs Sedentary Option
Other: Sedentary Option — Subjects will rate their liking of sedentary activities (reading magazines, playing word games, puzzles) as an alternative to exercise.

SUMMARY:
The purpose of this study is to understand how to make exercise more attractive to people.

DETAILED DESCRIPTION:
This investigation will address increased physical activity and will yield empirical evidence to inform developing tools to help individuals make healthy choices regarding physical activity (PA) and maintenance of healthy body weight. Behavioral Choice Theory provides a framework for understanding choices people make and how to shift an individual's choice toward healthier alternatives. The theory holds that choice is based on the relative motivating values of alternatives. One way to shift choice toward a healthier alternative is to increase the relative reinforcing value (RRV), or motivating value, of that alternative. Thus, increasing the RRV of PA behaviors could shift choice towards PA and away from less healthy, sedentary alternatives.

Increasing the RRV of PA may allow PA to compete with more reinforcing, sedentary behaviors, resulting in a shift in behavioral choice. This process is termed "incentive sensitization", which was originally proposed to explain drug addiction. Incentive Sensitization theory posits that the RRV of a behavior is increased through repeated exposures, which produce neuroadaptations that increase craving of the behavior - after repeated exposures to a stimulus, a 'sensitization' or hypersensitivity to the incentive motivational effects of the stimulus follows. Another factor that influences motivation for a behavior is the development of tolerance to unpleasant aspects of that behavior. Opponent-Process Theory would account for the acquisition of motives where the initial reinforcer may be negative - the affect experienced after repeated exposures is opposite to that experienced during the first few presentations. For exercise, this would include tolerance to any discomfort, pain, fatigue and displeasure and a greater positive post-exercise affective response: the affect experienced during and after exercise has a greater motivational significance in PA participation than knowledge and beliefs regarding health benefits. Therefore, the investigators propose that repeated exposures to PA will produce tolerance to unpleasant aspects while increasing the post-exercise affect. Sensitizing PA reinforcement and increasing discomfort tolerance may be associated with increasing the duration and intensity of daily activity. There are likely to be individual differences in sensitization of PA reinforcement and development of discomfort tolerance. Single-nucleotide polymorphisms (SNPs) that alter dopamine tone in the central dopaminergic reward system and SNPs associated with altered pain perception may contribute to such individual differences. The investigators anticipate that a moderate PA dose (300 kilocalorie [kcal] expenditure) will produce greater incentive sensitization and tolerance than a low dose (150 kcal) and that SNPs related to central dopamine tone and pain perception may contribute to individual differences in incentive sensitization and changes in physical activity after repeated exposures to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 19-35 kg/m2
* Healthy enough to exercise
* Sedentary (not regularly engaging in exercise more than once per week)

Exclusion Criteria:

* Taking any medications that affect energy expenditure or eating
* Have gained or lost more than 10 pounds over the past 3 months
* Use tobacco
* Pregnant or lactating or plan to become pregnant in the next 6 months
* Have any medical conditions that prevent the individual from safely joining in physical activity
* Have high work-related activity such as construction and farm work

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in relative reinforcing value (RRV) of physical activity | Week 0, Week 6, Week 10
  RRV of physical activity will be assessed by evaluating the number of responses (mouse button presses) a subject is willing to complete to gain access to physical activity or a sedentary alternative.
Changes in preference for intense physical activity and tolerance for exercise discomfort | Week 0, Week 6, Week 10
  Changes in preference for intense physical activity and tolerance for exercise discomfort will be assessed by self-report questionnaire responses to the Preference for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q).

SECONDARY OUTCOMES:
Change in minutes of physical activity, as assessed by activity tracker | Week 0, Week 6, Week 10
  Minutes of physical activity will be assessed by having participants wear an Actigraph accelerometer for 7 days (minimum 10 hours per day) on the right hip.
Changes in perceived support for physical activity from friends and family members | Week 0, Week 6, Week 10
  Changes perceived support for physical activity from friends and family members will be assessed by self-report questionnaire responses to the Social Norms and Support for Exercise Questionnaire.
Changes in perceptions of how much exercise satisfies autonomy, relatedness, and competence needs | Week 0, Week 6, Week 10
  Changes in perceptions of how much exercise satisfies autonomy, relatedness, and competence needs will be assessed by self-report questionnaire responses to the Psychological Need Satisfaction in Exercise Scale.
Changes in intrinsic, external, interrogated, identified, introjected and amotivation for physical activity | Week 0, Week 6, Week 10
  Changes in intrinsic, external, interrogated, identified, introjected and amotivation for physical activity will be assessed by self-report questionnaire responses to the Behavioral Regulation in Exercise, 3rd Edition (BREQ-3).
Changes in perceived effort expended during exercise | Week 0, Week 6, Week 10
  Changes in perceived effort expended during exercise will be assessed by self-report questionnaire responses to the Rating of Perceived Exertion Scale.
Changes in perceived pain/discomfort during exercise | Week 0, Week 6, Week 10
  Changes in perceived pain/discomfort during exercise will be assessed by self-report questionnaire responses to the Muscle Pain Questionnaire.
Changes in perceived ability to continue exercise long-term | Week 0, Week 6, Week 10
  Changes in perceived ability to continue exercise long-term will be assessed by self-report questionnaire responses to the Exercise Self-Efficacy Scale.
Changes in perceived ability to stick to an exercise routine | Week 0, Week 6, Week 10
  Changes in perceived ability to stick to an exercise routine will be assessed by self-report questionnaire responses to the Exercise Confidence Survey.
Changes in perceived affective responses to exercise | Week 0, Week 6, Week 10
  Changes in perceived affective responses (energy, tiredness, tension, calmness) to exercise will be assessed by self-report questionnaire responses to the Activation Deactivation Adjective Check List (ADCL).
Changes in average daily caloric intake | Week 0, Week 6, Week 10
  Changes in average daily calorie intake will be assessed by reporting all foods and beverages consumed over a 3-day period.

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No